CLINICAL TRIAL: NCT00417456
Title: The Development and Evaluation of an "E-Visit" Program for the Management of Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Director, Center for Connected Health, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2005-P-000289
Record Dates: First submitted 2006-12-29; First posted 2007-01-01 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Acne Vulgaris
Keywords: Acne; Telemedicine; Dermatology
MeSH Terms: conditions — Acne Vulgaris | interventions — Office Visits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Office Visits
  Interventions: Other: Office visit
- 2 (Experimental): Evisit
  Interventions: Other: Evisit

INTERVENTIONS:
Other: Evisit — Asynchronous,remote care delivery via a secure web platform
  Other Names: RelayHealth platform
  Arms: 2
Other: Office visit — Conventional office-based care
  Arms: 1

SUMMARY:
The purpose of this study is to test the efficacy, timeliness, and user satisfaction of an online "E-Visit" application that uses store-and-forward technology for acne patients requiring dermatologic care for their condition. Hypotheses:

1. That an "E-Visit" is an effective alternative to in-person clinic care for patients with mild to severe facial acne.
2. That providers and patients will be satisfied with this model.
3. That mean wait times for new and return visits will be reduced through the "E-Visit" model.
4. That this prototype for care will improve clinic workflow, offer additional patient access, and allow urgent cases to be seen earlier.

DETAILED DESCRIPTION:
Across the United States, a geographically mal-distributed workforce of Dermatologists exists, a problem that is projected to worsen. Patient access to dermatologic care is threatened. The dermatology workforce shortage has resulted in long wait times for patients, especially new patient visits and acute care cases.

Teledermatology has received much attention as a solution to the preceding problems. Teledermatology can reduce the burden of repeat office visits in chronic conditions by facilitating care from home. In this trial, a model incorporating store-and-forward technology is tested in general clinics while its impact on clinical outcomes, satisfaction, and wait times are studied.

Comparison: After consent, study subjects are assigned a unique study number and randomly assigned to one of two groups:

Group 1- The first group of subjects will have four (4) in-office visits spaced six weeks apart.

Group 2- The second group will have four (4) "e-visits" spaced six weeks apart.

At the end of study (after completion of 5th visit overall) all participants will complete a satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 or older
* Diagnosis of mild to severe facial acne
* Access to a credit card
* Access to an Internet connection and a computer
* Ability to image self
* MA Blue Cross/ Blue Shield Coverage

Exclusion Criteria:

* Non-English speaking individuals
* Patients taking Accutane for their acne
* Impaired Physical ability to image self
* Impaired Cognitive ability

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Peer review of subject images using the Total Inflammatory Lesion Count at the end of active recruitment | 6 months

SECONDARY OUTCOMES:
Subject satisfaction | 6 months
Physician satisfaction | 6 months
Timing of visits | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Kvedar, M.D., Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - MGH Dermatology Associates, Boston, Massachusetts
  - Brigham and Women's Hospital Department of Dermatology, Boston, Massachusetts

REFERENCES:
- [Derived] Watson AJ, Bergman H, Williams CM, Kvedar JC. A randomized trial to evaluate the efficacy of online follow-up visits in the management of acne. Arch Dermatol. 2010 Apr;146(4):406-11. doi: 10.1001/archdermatol.2010.29. PMID 20404229